CLINICAL TRIAL: NCT03419650
Title: Clinical Impact of Acthar in the Psoriatic Arthritis Patient (CLIPS)
Acronym: CLIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRIS Research and Development, LLC (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Guillermo Valenzuela, MD, Rheumatologist, IRIS Research and Development, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC0014
Record Dates: First submitted 2017-11-14; First posted 2018-02-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Psoriatic Arthritis
Keywords: PsA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Intervention Model Description: treatment arm will then be observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Other): treatment arm for 12 weeks followed by observation period of 12 weeks, and a bone density at week 52.
  Interventions: Drug: ACTHar

INTERVENTIONS:
Drug: ACTHar — Acthar™ 80 units twice a week for 4 weeks followed by 40 units twice a week until week 12.
  Other Names: acthar gel

SUMMARY:
Demonstrate the clinical value of Acthar TM in patients with active Psoriatic Arthritis who lack adequate response to DMARDS, and the quantification of response by clinical, serologic and structural parameters.

DETAILED DESCRIPTION:
The study is an investigator initiated study (IIS) single arm treatment, single center where patients will receive active treatment with ActharTM 80 units twice weekly for 4 weeks followed by 40 units twice weekly until week 12.

2-End points:

1.Primary Clinical Endpoint

1. To demonstrate the efficacy of Acthar for the treatment of patients with active psoriatic arthritis and who have not had an adequate response to non-biological DMARDs based on the proportion of subjects achieving a 20% improvement in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, Health Assessment Questionnaire (HAQ), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP) as described by American College of Rheumatology (ACR) 20 at week 12.

[Time Frame: 12 weeks]

2.Primary Imaging Endpoints

1. The improvement of the total DEMRIQ*-Volume score of synovial inflammation measured in the Metacarpophalangeal (MCP), proximal interphalangeal (PIP) and the distal interphalangeal (DIP) joints. [Time Frame: baseline to week 24]

   [Time Frame: baseline to week 24]
2. Secondary Outcome Measures:

Secondary Imaging Endpoints

1. The improvement in PSAMRIS* Synovitis score in the Metacarpophalangeal (MCP), proximal interphalangeal (PIP) and the distal interphalangeal (DIP) joints. [Time Frame: baseline to week 24]

[Time Frame: baseline to week 24]

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before any study-related procedure is undertaken that is not part of the standard subject management
2. Subjects are willing to comply with the structure of the study, such as visits, treatment plan, laboratory and imaging studies.

   Clinical evidence of psoriatic arthritis defined by at least 6 months of CASPAR defined criteria (evidence of current psoriasis, a personal history of psoriasis, or a family history of psoriasis. Current psoriasis is defined as psoriatic skin or scalp disease present today as judged by a rheumatologist or dermatologist. A personal history of psoriasis is defined as a history of psoriasis that may be obtained from a patient, family physician, dermatologist, rheumatologist, or other qualified health care provider. A family history of psoriasis is defined as a history of psoriasis in a first- or second-degree relative according to patient report, and the number of tender and swollen joints as later specified. Typical psoriatic nail dystrophy including onycholysis, pitting, and hyperkeratosis observed on current physical examination.

   c. A negative test result for the presence of rheumatoid factor by any method, according to the local laboratory reference range.

   d. Either current dactylitis, defined as swelling of an entire digit, or a history of dactylitis recorded by a rheumatologist.

   e. Radiographic evidence of juxtaarticular new bone formation, appearing as ill-defined ossification near joint margins (but excluding osteophyte formation) on plain radiographs of the hand or foot.

   Current psoriasis is assigned a score of 2; all other features are assigned a score of 1.

   The subject must have active arthritis at both screening and baseline, as defined by having both:
   * Tender/painful joints on motion (out of 68 joints assessed); and;
   * Swollen joints (out of 66 joints assessed). The subject must have active Plaque Psoriasis, which has been diagnosed, or confirmed by a rheumatologist or dermatologist and the ability to use skin biopsy as a diagnostic method.
3. Previous use of DMARDS:

   The practices for the administration of DMARD therapy, including laboratory testing, contraceptive requirements, follow-up care and contraindications should be performed according to local standards of care such as the ACR recommendations for monitoring for the duration of the study. Subjects should remain on a stable dose of that traditional DMARD throughout the course of the study.

   Methotrexate: Maximum dose of 15 mg/week. Minimum duration of therapy 3 months and dose stable for 4 weeks prior to first dose of the study. Subjects on methotrexate should be on an adequate and stable dose of folate supplementation.

   Sulfasalazine: Maximum dose of 3 gm/day. Minimum duration of therapy 2 months and dose stable for 4 weeks prior to first dose of study drug.

   Leflunomide: Maximum dose of 20 mg/day. Minimum duration of therapy 4 months and dose stable for 4 weeks prior to first dose of study drug.

   Plaquenil Azathioprine
4. Concomitant treatments:

   Corticosteroids up to 10 mg/day prednisone or prednisone equivalent are allowed for 4 weeks stable dose before the study and can be tapered according to the investigator criteria of clinical response. NSAIDS and COX 2 medications can be used in clinically accepted doses and in stable doses 4 weeks prior to screening. Topical keratolytics such as corticosteroids, tars, anthralin, vitamin D analogs, and retinoids must be discontinued 2 weeks prior to the screening date. Non-medicated emollients including 1% hydrocortisone for palms and soles are allowed. UV light therapy needs to be discontinued 2 weeks prior to screening, and PUVA 4 weeks prior to screening.
5. A male participant must agree to use and to have their female partners use a highly effective form of contraception, one day before the first dose of study treatment (as appropriate), during the treatment period, and refrain from donating sperm during this period.
6. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: age related amenorrhea for at least one year, and increased follicle-stimulating hormone (FSH) >40 Miu/Ml or who have undergone hysterectomy or bilateral oophorectomy are exempt from pregnancy testing.

A woman of childbearing potential is defined as a female capable of becoming pregnant. It is also defined as any female who has experienced menarche and is not permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without alternative medical cause.

Women of childbearing potential must agree to at least one method of birth control: a barrier method together or alone with a highly effective method to prevent pregnancy four weeks prior to randomization, throughout the study.

The definition of highly effective contraception includes:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; oral, intravaginal or transdermal,
* Progestogen-only hormonal contraception associated with inhibition of ovulation; oral, injectable or implantable,
* Intrauterine device,
* Intrauterine hormone-releasing system,
* Bilateral tubal occlusion,
* Vasectomized partner, or
* Sexual abstinence. b. Supplementary barrier methods include:
* Male or female condom with or without spermicide, or
* Cap, diaphragm or sponge with spermicide, c. Men must agree to use and have their female partners use a barrier method together with a highly effective contraceptive method as defined above.

Exclusion Criteria:

1. Other forms of psoriasis than plaque psoriasis.
2. Any person in direct relation to the study site such as employees or family members.
3. Breast feeding females, pregnant females or women in childbearing age not using adequate contraception.
4. Subjects participating in other concomitant investigational protocols.
5. Concurrent forms of severe, progressive disease such as renal, hepatic, hematological, gastrointestinal, pulmonary, neurologic and metabolic.
6. Blood cell count below 9g/dl of hemoglobin, wbc count of less than 3000/cubic millimeters, neutropenia of less than 1500/cubic millimeter, platelet count below 100,000/cubic millimeter.
7. Creatinine clearance of less than 40ml/min
8. Total bilirubin or transaminases 1.5 the normal value.
9. Known immunodeficiency
10. Subjects with other known autoimmune rheumatic disorder such as (Systemic Lupus Erythematosus (SLE), Mixed Connective Tissue Disease (MCTD)), or other known inflammatory disorders like gout, Lyme disease, infectious disorders.
11. History of Infected prosthesis
12. History of lymphoprolipherative disorder
13. History of recurrent disseminated herpetic infections.
14. Active infections, recent hospitalization for a condition requiring intravenous antibiotics, for three months since discharge.
15. Any form of biologic agent or patients who are active on chemotherapy or chemotherapy or any biologic within 6 months of the last treatment dose.
16. Alcohol abuse unless documented remission for more than 6 months
17. Acute psychiatric disorders or conditions that can alter the judgment of the subject.
18. Active Hepatitis B, and/or Hepatitis C.
19. Within one month prior to Screening, vaccination with live or live-attenuated virus vaccine.
20. Allergy to porcine derived substances, participants with congestive heart failure, and with osteoporosis are also excluded from the trial.

MRI related exclusion criteria In addition to the subjects matching the inclusion/exclusion criteria above, patients meeting any of the below must be excluded from the study.

* Known allergy to gadolinium or any of the excipients contained in the MRI contrast agent
* History of allergy
* Any metal objects e.g. Shrapnel, any surgical clips, pacemakers, pins, plates, screws, metal sutures or wire mesh also including uterine coil.
* Claustrophobia
* Morbid Obesity (BMI > 40kg/m2)
* Cochlear implants Caution is required for patients with tattoos: the patient should inform the MRI technician site staff, who will then be able to assess whether it is sage for the patient to undergo the MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Primary Clinical Endpoint | 12 weeks
  1. To demonstrate the efficacy of Acthar for the treatment of patients with active psoriatic arthritis and who have not had an adequate response to non-biological DMARDs based on the proportion of subjects achieving a 20% improvement in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, Health Assessment Questionnaire (HAQ), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP) as described by American College of Rheumatology (ACR) 20 at week 12.
Primary Imaging Endpoints | baseline to week 24
  1. The improvement of the total DEMRIQ*-Volume score of synovial inflammation measured in the Metacarpophalangeal (MCP), proximal interphalangeal (PIP) and the distal interphalangeal (DIP) joints. [Time Frame: baseline to week 24]

SECONDARY OUTCOMES:
Secondary Imaging Endpoints | baseline to week 24
  1. The improvement in PSAMRIS* Synovitis score in the Metacarpophalangeal (MCP), proximal interphalangeal (PIP) and the distal interphalangeal (DIP) joints. [Time Frame: baseline to week 24]

CONTACTS AND LOCATIONS:
Locations (1):
- IRIS Research and Development, Plantation, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided